CLINICAL TRIAL: NCT06085196
Title: Evaluation of an Outdoor Mindful Walking Program for Sustaining Cognitive Function in Older African Americans at Risk for Dementia
Brief Title: Mindful Walking Program for Older African Americans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chih-Hsiang Yang, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00123487
Record Dates: First submitted 2023-10-08; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Function; Aging Well; Behavior, Health
Keywords: Walking; Mindfulness; Lifestyle activity
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful walking (Experimental): Complete a 24-session outdoor mindful walking intervention over 3 months
  Interventions: Behavioral: Mindful walking activity
- Delayed mindful walking group (Other): Option to complete a delayed 24-session mindful walking
  Interventions: Behavioral: Mindful walking activity

INTERVENTIONS:
Behavioral: Mindful walking activity — Participate in 24 sessions of outdoor mindful walking on a local walking trail over three months

SUMMARY:
The goal of this clinical trial is to understand the beneficial role of mindful walking in sustaining cognitive health in African American older adults who have elevated risk of developing neuropsychological diseases. The main question it aims to answer is "Does a multi-session mindful walking intervention lead to promising signals of sustaining cognitive health in vulnerable AA older adults?" The researchers in this 2-arm randomized controlled trial will compare the mindful walking group with a delayed mindful walking to see if the intervention efficacy is observed at multiple follow-up period.

DETAILED DESCRIPTION:
African American (AA) older adults in the U.S. are disproportionally impacted by ADRD compared to other races and ethnicities. Mindful walking integrates two potentially protective factors of ADRD by elevating mindfulness and physical activity (i.e., walking), resulting in a synergistic behavioral strategy that is feasible and safe for older adults. However, the efficacy of using this intervention for cognitive health outcomes has not been tested using experimental designs. This study is a community-based, mindful walking randomized controlled trial to examine its efficacy on cognitive and other health outcomes in ADRD at-risk, AA older adults. This study will recruit 114 older adults (ages 60+ years) with elevated risk of developing ADRD from the Midlands region of South Carolina. Older adults were randomly assigned to participate in 24 sessions of mindful walking or a delayed mindful walking group (n=57 in each group). The study outcomes include various key brain health determinants, including cognitive function, quality of life, psychological well-being, physical activity, mindfulness, sleep, and overall health status. Participants in both groups follow identical measurement protocol of at baseline, 12 weeks, 18 weeks, and 24 weeks. The outcome measures are administered in the lab and in everyday settings. This study will generate preliminary evidence regarding the effects of mindful walking on sustaining cognition health. It will also inform future large-scale effectiveness trials to validate our study findings. If successful, this mindful walking program can be scaled up as a low-cost and viable lifestyle strategy to promote healthy cognitive aging in diverse older adult populations, including those at greatest risk.

ELIGIBILITY:
Inclusion Criteria:

1. African American ages 60 and above
2. Mild symptoms of cognitive decline or MCI
3. Physically inactive or insufficiently active (based on the 2018 US guidelines)
4. Adequate hearing and visual ability to complete study tasks and assessments
5. English proficiency
6. Medically stable with or without medication
7. Capable of providing informed consent
8. Willing to be randomized to one of the two groups

Exclusion Criteria:

1. Clinical diagnosis of ADRD or other brain abnormalities (e.g., strokes, epilepsy, Parkinson's disease
2. Clinical diagnosis of psychiatric disorders (i.e., depression, post-traumatic stress disorder, bipolar disorder)
3. Unable to walk independently (i.e., need caregiver's assistance) 4) Plan to have surgery or relocate outside the area within the next 6 months

5) Currently participate in other studies involving physical activity, mindfulness, or cognitive training

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function as assessed by the Montreal Cognitive Assessment (MoCA) | Baseline, 12,18,24 weeks follow-up
  MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, conceptual thinking, calculations, and orientation.
Everyday Cognition as assessed by the NIH Mobile Toolbox | Baseline, 18, 24 weeks follow-up (4 days each), Weeks 12 and 13 (14 days)
  The NIH Mobile Toolbox is a smartphone-based, ultra-brief cognitive assessments to measure different domains of cognition using the smartphone screen.

SECONDARY OUTCOMES:
Perceived Quality of Life as assessed by the EuroQol 5 dimensions and 5 levels questionnaire | Baseline, 12,18,24 weeks follow-up
  The EuroQol 5 dimensions and 5 levels survey (EQ-5D-5L) is a self-assessed, health related, quality of life questionnaire. The questionnaire measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, ranging from 11111 (best) to 55555 (worst).
Subjective Physical Activity Levels as assessed by the CHAMPS (Community Health Activities Model Program for Seniors) questionnaire | Baseline, 12,18,24 weeks follow-up
  The CHAMPS self-report questionnaire assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults
Device-based Physical Activity Levels as assessed by the activPAL Accelerometer | Weeks 12 and 13 (14 days)
  The activPAL is a small, slim activity monitor that uses an accelerometer to measure limb position and activity. It's worn on the thigh and uses algorithms to determine body posture, including moving, standing, and sitting.
Mindfulness Level as assessed by the Mindfulness Attention Awareness Scale and Five Facet Mindfulness Questionnaire | Baseline, 12,18,24 weeks follow-up
  Use Mindfulness Attention Awareness Scale (MAAS) is a 15-item self-report survey that measures mindfulness in general and in specific day-to-day circumstances. Each MAAS scores can range from 1 to 6. Higher scores indicate greater mindfulness; The Five Facet Mindfulness Questionnaire (FFMQ) has 39 self-reported items. It measures five mindfulness facets, including Observing, Describing, Acting with awareness, Non-judgmental, and Non-reactive. The items are rated on a 5-point Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true).
Overall Health Status as assessed by the SF-36 self-report survey | Baseline, 12,18,24 weeks follow-up
  The SF-36 is a 36-item survey that measures eight domains of health status. The survey is designed to capture adult patients' perceptions of their own health and well-being. The score range is 0 to 100. Higher scores indicate better health status.
Mobility as assessed by the 10-meter walk test | Baseline, 12,18,24 weeks follow-up
  The 10-meter walk test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
Perceived Stress as assessed by the Perceived Stress Scale (PSS-10) | Baseline, 12,18,24 weeks follow-up
  The Perceived Stress Scale (PSS-10) is a 10-item questionnaire that measures psychological stress. The PSS-10 asks respondents to rate statements about their feelings and thoughts. Each question is scored from 0 (never) to 5 (very often) with a total possible score range of 0 to 40.
Depressive Symptoms as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, 12,18,24 weeks follow-up
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a 20-item questionnaire that measures the severity of depressive symptoms in the general population. The CES-D has a possible range of scores from zero to 60. Higher scores indicate the presence of more symptomatology.
Sleep Quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 12,18,24 weeks follow-up
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire that assesses sleep quality and quantity. It has seven components, each rated from 0 (no difficulty) to 3 (severe difficulty). It has a global score range of 0 to 21. Higher scores indicate worse sleep quality.

OTHER OUTCOMES:
Height as measured from the top of the person's head to the heel using digital stadiometer | Baseline
  Use the PhenX Toolkit protocol and measure height in duplicates. The height measurements is taken to the nearest 0.1 cm. A third measurement is conducted if the first two measurements differ by more than 1.0 cm.
Weight as measured using a digital floor scale | Baseline
  Use the PhenX Toolkit protocol and measure weight in duplicates. The weight measure is conducted to the nearest 100 grams. If the first two measurements differ by more than 200 grams or 0.25 pounds, a third measurement should be taken.
Body Mass Index (BMI) as calculated by the height and weight measures | Baseline
  Body mass index (BMI) is a value derived from the mass and height of a person. The BMI is defined as the body mass divided by the square of the body height. Major adult BMI classifications are underweight (under 18.5 kg/m2), normal weight (18.5 to 24.9), overweight (25 to 29.9), and obese (30 or more).
Waist Circumference as measured using a tape measure at the uppermost lateral border of the ilium | Baseline
  Waist circumference is a more direct measure of central obesity. It's a marker for visceral fat, which plays a role in the development of many chronic diseases, including type 2 diabetes and cardiovascular disease.
Systolic and diastolic blood pressures as measured using the automatic arm blood pressure monitor | Baseline
  Blood pressure is the pressure, measured in millimeters of mercury, within the major arterial system of the body. It is conventionally separated into systolic and diastolic determinations. Systolic pressure is the maximum blood pressure during contraction of the ventricles; diastolic pressure is the minimum pressure recorded just prior to the next contraction.
Health Literacy as assessed by a validated survey item | Baseline
  Use one valid item from the Wallace et al. (2006) publication - Screening Items to Identify Patients with Limited Health Literacy Skills. The study concluded that a single question is sufficient to identify patients with limited health literacy.
Grip Strength as measured using the digital dynamometer | Baseline
  This dynamometer is designed for home, sport, and clinical use to measure grip strength. It has a high precision power gauging that gives an accurate digital reading of gripping power. The handle can be adjusted up or down to get an ideal grasp.
Daily Functioning as assessed by the Brody Instrumental Activities of Daily Living Scale (IADL) | Baseline
  The Lawton Instrumental Activities of Daily Living (IADL) Scale assesses a person's ability to perform daily living tasks. The scale measures eight domains, including: Using the telephone, Shopping, Food preparation, Housekeeping, Laundry, Transport, Medication, Finances. The scale has eight items and takes about 10 to 15 minutes to administer. The summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
Social Support as assess by the Perceived Social Support Scale (PSSS) | Baseline
  PSSS is a 12-item questionnaire that uses a 7-level scoring method (from 1 = "disagree" to 7 = "extremely agree"). The total score ranges from 12 to 84 points. Higher scores indicate a higher level of the individual's perception of social support.
Medication Use as assessed using the general health needs survey | Baseline
  The general health needs survey question was developed and validated in 2014 by the UnitedHealthcare to screen for health status. The survey asks respondents if they used prescription drugs for any reason in the past 12 months or lifetime and what are the prescription drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsiang "Jason" Yang, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Yang CH, Lee J, Wilcox S, Rudisill AC, Friedman DB, Hakun JG, Neils-Strunjas J, Wei J, Miller MC, Byers MD. Implementation and evaluation of a community-based mindful walking randomized controlled trial to sustain cognitive health in older African Americans at risk for dementia. BMC Geriatr. 2024 Jul 4;24(1):579. doi: 10.1186/s12877-024-05090-2. PMID 38965464